CLINICAL TRIAL: NCT05760989
Title: Edwards EWJ-202 Transcatheter Tricuspid Valve Replacement System: Investigation of Safety and Clinical Efficacy Using a Novel Device in Patients With at Least Severe Tricuspid Regurgitation in JAPAN
Brief Title: TRISCEND JAPAN Study
Acronym: TRISCEND JAPAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Tricuspid Valve Regurgitation; Heart Valve Diseases; Cardiovascular Diseases
Keywords: Transcatheter; Tricuspid Disease; Valve Replacement; Tricuspid Valve
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with the Edwards EWJ-202 Transcatheter Tricuspid Valve Replacement System (Experimental)
  Interventions: Device: Edwards EWJ-202 Transcatheter Tricuspid Valve Replacement System

INTERVENTIONS:
Device: Edwards EWJ-202 Transcatheter Tricuspid Valve Replacement System — Replacement of the native tricuspid valve through a transcatheter approach

SUMMARY:
A prospective, open, non-randomized, multicenter, clinical trial to evaluate the safety and effectiveness of the Edwards EWJ-202 transcatheter tricuspid valve replacement system in the treatment of patients with at least severe tricuspid regurgitation despite medical therapy. Subjects will be followed at discharge, 30 days, 6 months and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic tricuspid regurgitation (TR) despite medical therapy
* TR graded as severe or greater
* Appropriate for transcatheter tricuspid valve replacement per the local heart team

Exclusion Criteria:

* Tricuspid valve anatomic contraindications
* Need for emergent or urgent surgery or any planned cardiac surgery within the next 12 months
* Hemodynamic instability
* Refractory heart failure requiring advanced intervention
* Currently participating in another investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | 1 year
  Participants with all-cause mortality at 1 year from the index procedure
Heart Failure Hospitalization | 1 year
  Participants with a heart failure hospitalization at 1 year from the index procedure

SECONDARY OUTCOMES:
Rates of various adverse events | 30 days, 6 months, 12 months, annual for five years
  Rates of various adverse events as defined in the protocol
Rate of Major Adverse Events (MAEs) | 30 days
  Composite rate of MAEs as defined in the protocol
Reduction in TR grade | 30 days, 6 months, 12 months, annual for five years
  Number of participants with reduction in TR from baseline
New York Heart Association (NYHA) Functional Class | 30 days, 6 months, 12 months, annual for five years
  Number of participants with improvement in NYHA class
Health Status as measured by the SF-36 Questionnaire | 30 days, 6 months, 12 months, annual for five years
  Number of points of improvement in health status as measured by 36-item short form survey (SF-36)
Health Status as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 30 days, 6 months, 12 months, annual for five years
  Number of points of improvement in health status as measured by KCCQ
Health Status as measured by the EQ-5D-5L Questionnaire | 30 days, 6 months, 12 months, annual for five years
  Number of points of improvement in health status as measured by EQ-5D-5L Questionnaire
Six-minute walk test | 30 days, 6 months, 12 months, annual for five years
  Change in distance (m) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiro Morino, MD, Study Chair — Iwate Medical University Hospital
Locations (8):
- Japan (8):
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Osaka Keisatsu Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No